CLINICAL TRIAL: NCT05776342
Title: Prognostic and Predictive Markers of Treatment Response in Patients With Pancreatic Adenocarcinoma
Brief Title: Prognostic and Predictive Markers of Treatment Response in Patients With PAC.
Acronym: CANOPE
Status: Recruiting | Type: Observational
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Other Study IDs: CANOPE GB-121
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to identify prognosis and predictive markers of response to treatments (surgery, chemotherapy,...) in patients with pancreatic adenocarcinoma. The effectiveness and tolerance of these treatments in current practice is also evaluated.

DETAILED DESCRIPTION:
The modest efficacy of current therapies for pancreatic cancer calls for the development of prognostic factors to guide patient selection and clinical decision-making based on tumor aggressiveness and risk of death.

The aim of this study is to identify prognostic and predictive factors of response to treatments administered in pancreatic adenocarcinoma, based on a multicenter cohort established on a population derived from current clinical practice. By accurately stratifying patients according to their estimated survival, prognostic tools could aid therapeutic decisions and optimize patient selection in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed pancreatic adenocarcinoma.
* Disease at a resectable, borderline, locally advanced, initially metastatic, or recurrent stage after surgery
* Diagnosis between January 1, 2003, and December 31, 2030.
* First-line treatment with chemotherapy and/or radiotherapy and/or clinical trials.
* Age ≥ 18 years.
* Written informed consent

Exclusion Criteria:

* Patient under guardianship, curatorship, or judicial protection.
* Pregnant or breastfeeding women.
* Any medical, psychological, or social situation that could prevent compliance with the protocol as assessed by the investigator.
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retro-prospective (diagnosis between 2003 and 2022) and prospective (diagnosis between 2023 and 2030) cohorts of patients with pancreatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 4050 (Estimated)
Dates: Start 2003-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) rate | Up to 7 years from the date of initial cancer diagnosis (or until death if it occurs before 17 years)
  Defined as the time interval between the start date of treatment (surgery, first cycle of L1 chemotherapy, or first radiotherapy session) and the date of death regardless of the cause. Living or lost to follow-up patients will be censored at the date of the last news

SECONDARY OUTCOMES:
Progression-free survival (PFS) rate | Up to 7 years
  Defined as the time interval between the start date of treatment (surgery, first cycle of L1 chemotherapy, or first radiotherapy session) and the date of first progression or date of death regardless of the cause. Living patients without progression or lost to follow-up will be censored at the date of the last news
Number of patient with objective response rate | Up to 7 years
  Evaluation according to RECIST v1.1, Choi or iRECIST criteria. Study the population followed for pancreatic adenocarcinoma according to tumor stages (localized, borderline, locally advanced, metastatic or recurrent after surgery) and according to treatments.
Number of patient with stability rate | Up to 7 years
  Evaluation according to RECIST v1.1, Choi or iRECIST criteria. Study the population followed for pancreatic adenocarcinoma according to tumor stages (localized, borderline, locally advanced, metastatic or recurrent after surgery) and according to treatments.
Number of patient with tumor progression | Up to 7 years
  Evaluation according to RECIST v1.1, Choi or iRECIST criteria. Study the population followed for pancreatic adenocarcinoma according to tumor stages (localized, borderline, locally advanced, metastatic or recurrent after surgery) and according to treatments.
Number of patient with grade 3/4 treatment-related toxicities | Up to 7 years
  Toxicity rates according to CTCAE v5.0 classification. Study the population followed for pancreatic adenocarcinoma according to tumor stages (localized, borderline, locally advanced, metastatic or recurrent after surgery) and according to treatments.
Number of patients who received maintenance treatment in the first-line | Up to 7 years
  Study the profiles of patients receiving maintenance treatment in 1st-line chemotherapy
Number of patients who received second and third-line treatments | Up to 7 years
  Study the profiles of patients receiving 2nd and 3rd lines of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Angelique VIENOT, MD, Principal Investigator — CHRU de Besançon - Institut Régional Fédératif du Cancer (IRFC) de Franche-Comté; Anthony Turpin, MD, Principal Investigator — Hôpital Claude-Huriez
Locations (15):
- France (15):
  - CHU Jean Minjoz, Besançon
  - Hôpital Beaujon, Clichy
  - CHU - Henri Mondor, Créteil
  - CHU Lille, Lille
  - Centre Léon Bérard, Lyon
  - HRU Nancy Site Brabois, Nancy
  - Hôpital Georges Pompidou, Paris
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Pontchaillou, Rennes
  - Institut Curie, Saint-Cloud
  - IHU - Institut de chirurgie guidée par l'imagerie, Strasbourg
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No